CLINICAL TRIAL: NCT01527305
Title: An Open-Label, Prospective, Non-Comparative Study to Evaluate the Efficacy and Safety of Paliperidone Palmitate in Subjects With Acute Schizophrenia
Brief Title: A Study to Evaluate the Effectiveness and Safety of Paliperidone Palmitate in Subjects With Acute Schizophrenia
Acronym: PREVAIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100739; R092670SCH4009 (Other: Johnson & Johnson Pte Ltd.); PALM-KOR-4004 (Other: Johnson & Johnson Pte Ltd.); PALM-KOR-4003 (Other: Johnson & Johnson Pte Ltd.)
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotics; Paliperidone Palmitate; Paliperidone; Invega; Sustenna; Psychotic disorder; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Paliperidone palmitate (Experimental)
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate — Participants will receive 1 intramuscular (into muscle) injection of 150 milligram (mg) on Day 1 and 1 injection of 100 mg on Day 8. Participants will also receive the last 2 paliperidone intramuscular injections between 50 - 150 mg (based on effectiveness and safety profile), on Day 36 and Day 64.
  Other Names: Sustenna

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of paliperidone palmitate in schizophrenic inpatients who have experienced recent exacerbation of acute schizophrenia (that is within past 4 weeks).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (looking forward using periodic observations collected predominantly following participant enrollment), non-comparative and multicenter study to evaluate the effectiveness and safety of paliperidone palmitate in acute schizophrenic participants. This study consists of a screening phase (up to 7 days), treatment phase (13 weeks), and a study completion or early withdrawal visit. Safety evaluations will include adverse events, clinical laboratory tests, concomitant medications, physical examination, and vital signs, which will be monitored throughout the study. The total duration of study participation for each participant will be approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders Version IV (DSM-IV)
* Must be admitted to a hospital within 4 weeks prior to Screening experiencing an acute exacerbation of schizophrenia
* Have a positive and negative syndrome scale (PANSS) total score of more than or equal to 60 or clinical global impressions - severity (CGI-S) score of more than or equal to 4 (moderately ill) at Screening
* Agree to protocol-defined method of contraception
* Must be medically stable based on physical examination, medical history, vital signs, and clinical laboratory tests performed at Screening

Exclusion Criteria:

* Have a primary active DSM-IV Axis I diagnosis other than schizophrenia
* Have evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal, neurological, endocrine, metabolic or pulmonary disease in medical history, clinical laboratory or physical examination
* Have a history of neuroleptic malignant syndrome
* Participants at risk of suicide
* Have received clozapine within 1 month prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-06-22 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score | Baseline (Week 0), Week 13
  The PANSS is scale of 30 items which includes 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items). Each item is rated on a scale of 1 (absent) to 7 (extreme). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).

SECONDARY OUTCOMES:
Number of Participants With at Least a 30 Percent Reduction From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score | Baseline, Week 13
  The PANSS is scale of 30 items which includes 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items). Each item is rated on a scale of 1 (absent) to 7 (extreme). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Factor Scores | Baseline, Week 13
  Marder factor scores of the PANSS, derived by factor-analysis includes 5 factors: negative symptom, positive symptom, disorganized thought, uncontrolled hostility/excitement, and anxiety/depression factor scales. Positive factor score (range: 8 to 56): sum of select scores from positive, negative, and general psychopathology subscales. Negative factor score (range: 7 to 49): sum of select scores from negative and general psychopathology subscales. Disorganized thoughts factor score (range: 7 to 49): sum of select scores from positive, negative, and general psychopathology subscales. Uncontrolled hostility/excitement factor score (range: 4 to 28): sum of select scores from positive and general psychopathology subscales. Anxiety/Depression factor score (range: 4 to 28): sum of select scores from general psychopathology subscale. Higher scores indicate worsening.
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Subscale Scores | Baseline, Week 13
  The PANSS is scale of 30 items which includes 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items). The scale ranges from 1 (absent) to 7 (extreme). Each item is rated on a scale of 1 (absent) to 7 (extreme). The subscale score is the sum of scores of items in the subscale. Positive subscale (range: 7 to 49), negative subscale (range: 7 to 49) and general psychopathology subscale (range: 16 to 112). Higher scores indicate worsening.
Change From Baseline in Global Severity of Illness Using the Clinical Global Impression - Severity (CGI-S) Score | Baseline, Week 13
  The CGI-S rating scale is used to rate the severity of a participant's overall clinical condition on a 7-point scale ranging from 1 to 7 where 1=Normal, not at all ill, 2=Borderline mentally ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, 7=Among the most extremely ill.
Change From Baseline in Personal and Social Performance (PSP) Scale Score | Baseline, Week 13
  The PSP assesses the overall personal and social functioning on a continuum from grossly impaired functioning to excellent functioning using 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The degree of dysfunction a participant exhibits during the month prior to the assessment is rated on a 6-point scale (1=absent, 2=mild, 3=manifest, 4=marked, 5=severe, 6=very severe). The final total score ranges from 1 - 100 (71 - 100 indicating mild, good or excellent degree of dysfunction, 31 - 70 indicating varying degrees of difficulty, and <=30 indicating such a poor level functioning that intensive supervision is required).
Time to Readiness for Hospitalization Discharge for Inpatients Using the Readiness for Discharge Questionnaire (RDQ) Scale | Baseline up to Week 13
  The 6-item RDQ consists of 5 items assessing suicidality/homicidality, control of aggression/impulsivity, activities of daily living, independence in medication-taking, delusions/hallucinations interfering with functioning, on a 4-point scale (1=strongly agree, 2=agree, 3=disagree, 4=strongly disagree), and 1 item assessing CGI-severity <=4 status using a binary (yes/no) response. Using all 6 items as a guide, the clinician provides a final overall "yes/no" answer to the question 'is the participant ready for discharge'.
Number of Participants With Drug Discontinuation | Up to Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- China (6):
  - Huzhou
  - Shanghai
  - Shantou
  - Suzhou
  - Wenzhou
  - Wuxi
- Malaysia (3):
  - Johor Bahru
  - Kuala Lumpur
  - Tanjong Rambutan
- South Korea (7):
  - Busan
  - Goyang
  - Gyeonggi-do
  - Jeonju
  - Kyounggi
  - Seoul
  - Suwon
- Taiwan (5):
  - Douliou City, Yunlin County
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei

REFERENCES:
- See also: An Open-label, Prospective, Non-comparative Study to Evaluate the Efficacy and Safety of Paliperidone Palmitate in Subjects with Acute Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3404&filename=CR100739_CSR.pdf